CLINICAL TRIAL: NCT03978897
Title: A Randomized Controlled Trial of Blood Flow Restriction Plus Conventional Physical Therapy vs. Conventional Physical Therapy Alone in the Treatment of Lateral Epicondylitis
Brief Title: Trial of Blood Flow Restriction Plus Physical Therapy vs. Physical Therapy Alone for Lateral Epicondylitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Akron General (Other)
Responsible Party: Principal Investigator, Aaron Lear, Director of Primary Care Sports Medicine, Cleveland Clinic Akron General
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19001
Record Dates: First submitted 2019-05-24; First posted 2019-06-07 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; tennis elbow; blood flow restriction; physical therapy
MeSH Terms: conditions — Tennis Elbow | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Treating therapists and patient will be aware of treatment. The outcome assessor will have access to outcome data only, without knowledge of which treatment patient received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Blood flow restriction with physical/occupational therapy (Experimental): physical/occupational therapy including use of blood flow restriction tourniquet over 6 visits (within a twelve week period).
  Interventions: Device: Blood flow restriction tourniquet
- Evidence based physical/occupational therapy (Active Comparator): evidence based physical/occupational therapy program over 6 visits (within a twelve week period) without use of blood flow restriction tourniquet
  Interventions: Other: Evidence based physical/occupational therapy

INTERVENTIONS:
Device: Blood flow restriction tourniquet — A blood flow restriction tourniquet, which impedes arterial flow to extremity at 50% of usual flow.
  Other Names: Delfi personalized tourniquet system
  Arms: Blood flow restriction with physical/occupational therapy
Other: Evidence based physical/occupational therapy — Up to date physical/occupational therapy for lateral epicondylitis
  Arms: Evidence based physical/occupational therapy

SUMMARY:
Open label randomized controlled trial comparing evidenced based physical/occupational therapy vs. physical/occupational therapy including blood flow restriction tourniquet in the treatment of lateral epicondylitis (tennis elbow).

DETAILED DESCRIPTION:
Patients will be randomized to one of two groups, and treatment will be open label and unblinded. A target of 44 patients for enrollment has been set for 80% power. Treatment will last for 6 visits with physical therapy with recommended visit intervals of 1 week :

Intervention Group: Evidence based physical/occupational therapy, with the addition of therapeutic exercises using a blood flow restriction tourniquet.

Control Group: Patients will receive standard evidence based physical therapy

The primary outcome (Patient-Rated Tennis Elbow Evaluation [PRTEE]) will be collected at enrollment, 3, 6, and 12 months.

Secondary outcomes will be collected at the beginning and end of physical therapy interventions (change in: numeric pain rating scale, maximum pain free grip strength, pain free grip strength). We will collect treatments received after the end of physical therapy and before final follow up.

ELIGIBILITY:
Inclusion Criteria:

* The diagnoses included are lateral elbow pain, lateral epicondylitis, or lateral epicondylalgia, more general diagnoses elbow tendinitis or elbow pain will be included if their clinical picture at physical therapy meets criteria for lateral epicondylitis.
* If the inclusion diagnosis is other than lateral epicondylitis or tennis elbow (such as elbow pain), we will confirm the diagnosis at the first therapy visit with tenderness at the lateral epicondyle and/or pain with resisted wrist/long finger extension at the lateral epicondyle.
* Pain for 4 weeks or more.
* All participants must be between the age of 18 and 70 years old and have had pain for 4 weeks or more.

Exclusion Criteria:

* Ligamentous elbow sprain, osteoarthritis of elbow and cervical radiculopathy in the affected limb will be excluded from the study.
* Any history of ligamentous, bony or other soft tissue reconstruction surgery at the affected elbow,
* Vascular disorders to include: history of DVT, history of endothelial dysfunction, peripheral vascular disease
* Injection therapy (corticosteroid, platelet rich plasma, or other injection therapy) in the prior 3 months to the affected site
* Current fracture in affected arm
* History of crush injury to affected arm
* Any surgery on affected arm in last 1 year
* Surgical procedure on their contralateral extremity (Changed 9/2019 to surgery within last year on contralateral upper extremity).
* History of lymphectomy (such as axillary exploration with breast surgery, lymph node biopsy in the affected axilla/arm)
* Pregnancy
* Active infection
* Current cancer diagnosis/treatment
* Sickle cell anemia or trait
* Kidney dialysis
* History of syncope/passing out with pressure to body (such as massage, or blood pressure cuff).
* inability to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient rated tennis elbow evaluation (PRTEE) | 12 months
  Change in score on 'Patient rated tennis elbow evaluation' total score. Lower numbers suggest less pain, higher scores suggest more pain. Total score 0-100.
  Includes pain subscale (0-50)
  Specific activities subscale (0-60)
  Usual activities subscale (0-40)
  Function Subscale= (specific activities score + usual activities score)/2 (0-50)
  Total Score= Pain subscale + Function Subscale (0-100)

SECONDARY OUTCOMES:
Numeric pain rating scale | 12 months
  change in score on 0-10 pain rating scale with 0 being no pain, and 10 being worst pain.
Pain free grip strength | at final therapy visit up to 12 weeks after enrollment
  Change in pain free grip strength on dynamometer
Maximum grip strength | at final therapy visit up to 12 weeks after enrollment
  Change in maximum grip strength on dynamometer
Other treatments received | 12 months
  We will collect data on whether the patient sought or received treatments beyond physical/occupational therapy over the 12 months of enrollment in the study

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lear, MD, CAQ, Principal Investigator — Cleveland Clinic Akron General
Locations (1):
- Cleveland Clinic Akron General, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No